CLINICAL TRIAL: NCT01545648
Title: Pilot Study to Evaluate the Impact of Denosumab on Disseminated Tumor Cells (DTC) in Patients With Early Stage Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: Hope Rugo, MD (Other)
Collaborators: University of California, San Francisco (Other); Amgen (Industry)
Responsible Party: Sponsor-Investigator, Hope Rugo, MD, Clinical professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 117527; NCI-2012-02802 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2012-02-27; First posted 2012-03-07 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Early Stage Breast Cancer
Keywords: breast; cancer; early; DTC; disseminated; tumor; cells
MeSH Terms: conditions — Neoplasms | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- denosumab (Experimental): Dosage: 120 mg, monthly for total of 6 months, then every 12 weeks for 2 doses, for a total treatment course of one year
  Route of administration: subcutaneous injection
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab — Formulation of Dosage forms
  The vial presentations of denosumab contain 60 mg/mL denosumab, 17 mM sodium acetate, and 4.7% (w/v) sorbitol, at a pH of 5.2, filled to a target deliverable volume of 1.0 mL; or 70 mg/mL denosumab, 18 mM sodium acetate and 4.6% (w/v) sorbitol, at a pH of 5.2, filled to a target deliverable volume of 1.7 mL. The prefilled syringe (PFS) drug product contains denosumab at 60 mg/mL, 17 mM sodium acetate, 4.7% (w/v) sorbitol, and 0.01% (w/v) polysorbate 20, at a pH of 5.2, filled to a target deliverable volume of 1.0 mL.
  Dosage: 120 mg, monthly for total of 6 months, then every 12 weeks for 2 doses, for a total treatment course of one year
  Route of administration: subcutaneous injection
  Other Names: AMG 162; XGEVA™; Prolia®

SUMMARY:
The purpose of this study is to see whether taking denosumab for 12 months in women with a significant number of disseminated tumor cells in the bone marrow can reduce the number of these cells below a significant level.

DETAILED DESCRIPTION:
The presence of disseminated tumor cells (DTC) in the bone marrow in women with early stage breast cancer is an important prognostic factor associated with an increase in both recurrence and disease-associated death. In a pooled analysis of 4703 invasive breast cancer patients, detection of DTC in the bone marrow was associated with an increase in disease recurrence, distant metastases, and death from breast cancer over a median follow-up period of 5.2 years. Subsequent studies have demonstrated that the presence of DTC in the bone marrow of women with early breast cancer following completion of adjuvant therapy have an even greater impact on the risk of recurrence and death from breast cancer. Multivariate analysis demonstrated that the presence of marrow cells was an independent prognostic factor for reduced breast cancer specific survival with a relative risk of 6.3 (2.3-17.6, p<0.0001). Clearly, the detection of DTC in women with early stage breast cancer is a marker for increased risk of relapse and death, and this could serve as a unique indicator to select higher risk patients for intervention with targeted therapeutics.

It has long been recognized that there is close relationship between bone and immune system, recent studies also suggests that in addition to monocytes/macrophage, T cells (especially Th17, a subset of T helper cells that produces IL-17), B cells and dendritic cells all play an important role in osteoclast formation. RANKL, in addition to its effect on osteoclasts, also induces local inflammation. Several recent studies have demonstrated that the presence of tumor associate macrophages (TAM) is associated with more aggressive disease, and a worse outcome. Preclinical data suggests that TAM plays an important role in promoting metastases and resistance to therapy. In addition to RANKL, there are other genes secreted by breast cancer cells, including TGF-β, TNF associated factor 6 (TRAF6), Hypoxia Induced Factor -1 (HIF-1) and Bone morphogenetic protein 2 (BMP2), also involve in bone-cancer "vicious cycle" and induce RANKL expression. Cytokines, such as IL-4, IL-6, IL-17, TNF-α and CSF-1, also play an important role in osteolysis and immune response in bone microenvironment by regulating TAM function (CSF-1, IL-4 and IL-17) and RANKL expression. Recently, CD47 and Signal Regulatory Protein α (SIRPA) were also shown to impair macrophage function, and associated with increased risk for recurrence in patients with breast cancer. The investigators hypothesize that patients with higher DTC may have higher expression of RANKL and chronic inflammatory cytokines. The investigators plan to evaluate the expression of RANK, RANKL, TRAF6, BMP2, CSF-1, CD47, IL-17 and SIRPA on isolated DTC and bone marrow hematopoietic cells, and correlate these results to the outcome of patients enrolled in the trial.

The investigators hypothesize that treatment with denosumab will decrease the number of DTC in women with early stage breast cancer who have completed adjuvant or neoadjuvant cytotoxic therapy possibly by preventing cancer cell migration, and by promoting cancer cell death by changing the bone into a "hostile" environment .

The investigators propose to conduct a non-randomized phase II trial testing this hypothesis in women with early stage breast cancer and persistent DTC following adjuvant systemic therapy. Patients with DTC will receive denosumab monthly for 6 months, then every 3 months for a total of one-year treatment, to mirror the schedule utilized in the ongoing randomized phase III denosumab versus placebo D-CARE trial. DTC will be monitored following 6 months and 12 months of therapy. The investigators anticipate that this treatment will reverse the "vicious cycle" between bone and cancer cells.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years of age with histologically or cytologically confirmed stage I, II, or III breast cancer.
2. ECOG Performance Status of 0 or 1
3. Prior therapy:

   1. Prior adjuvant therapy is not required for participation in this study.
   2. If adjuvant or neoadjuvant treatment with chemotherapy is recommended, it must be completed before study start, and not more than 18 months prior to study start.
   3. If adjuvant or neoadjuvant treatment with trastuzumab (Herceptin®) is recommended, patients should have received at least 3 months of therapy before eligibility bone marrow is performed.
   4. Patients who have had surgery following neoadjuvant chemotherapy or hormonal therapy are eligible
   5. Patients must have completed definitive surgery and have completely resected disease.
   6. Concomitant hormonal therapy is allowed.
   7. Concomitant adjuvant trastuzumab is permitted
   8. If adjuvant hormonal treatment is recommended, patients should have received at least 3 months of therapy before screening bone marrow is performed.
4. Bone marrow aspirate positive by IE/FC assay within 12 weeks of study entry

   1. Definition of positive: >10 DTC/ml
   2. Timing of bone marrow aspiration to determine study eligibility

   i.If patient is to receive either no adjuvant therapy or hormonal therapy alone, the aspiration may be performed at diagnosis as part of the large micrometastasis study at UCSF, or following diagnosis if the patient received initial surgery elsewhere. This is also true for patients who have surgery following neoadjuvant therapy for breast cancer.

   ii.If the patient is to receive adjuvant chemotherapy, the aspiration will be performed at least three weeks after chemotherapy has been completed.

   iii.For trastuzumab and hormone therapy, see above.
5. Laboratory studies

   1. Liver function tests within normal limits, including total bilirubin, alkaline phosphatase, and AST (elevation of total bilirubin due to Gilbert's disease is allowed).

      * Gilbert's disease: a common hereditary cause of increased indirect bilirubin, but with normal direct bilirubin.
   2. Calculated creatinine clearance (calculated GFR) > 30 ml/min
6. Ability to understand and sign informed consent
7. Patients who have had surgery following neoadjuvant chemotherapy or hormonal therapy are eligible to participate in this trial.

Exclusion Criteria:

1. Karnofsky performance status < 90%
2. Patients participating in this study are not allowed to receive bisphosphonate therapy during the study period, either oral or intravenous.
3. Patients who completed adjuvant or neoadjuvant therapy more than 18 months prior to study screening.
4. A history of malignancy within the last 5 years except basal cell carcinoma of skin.
5. A history of human immunodeficiency virus (HIV) infection.
6. Severe, concurrent illness that would likely prevent the patient from being able to comply with the study protocol.
7. Pregnant or lactating women and women of child-bearing potential who are not using an effective method of birth control.
8. Significant dental disease that requires major intervention during the study period, such as tooth extraction
9. Significant coagulopathy that would prevent safe bone marrow aspiration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2015-06-09 (Actual); Study Completion 2016-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hope Rugo, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stefanovic S, Diel I, Sinn P, Englert S, Hennigs A, Mayer C, Schott S, Wallwiener M, Blumenstein M, Golatta M, Heil J, Rom J, Sohn C, Schneeweiss A, Schuetz F, Domschke C. Disseminated Tumor Cells in the Bone Marrow of Patients with Operable Primary Breast Cancer: Prognostic Impact in Immunophenotypic Subgroups and Clinical Implication for Bisphosphonate Treatment. Ann Surg Oncol. 2016 Mar;23(3):757-66. doi: 10.1245/s10434-015-4895-3. Epub 2015 Oct 14. PMID 26467455

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Patients will be treated with denosumab at a dose of 120 mg by subcutaneous injection monthly(-3/+3 days) for total of 6 months, then every 12 weeks (-7/+7 days) for 2 doses, for a total treatment course of one year.
Period: Overall Study
Arm/Group | Treatment
Started | 4
6 Months of Treatment | 4
Completed (12 months of treatment) | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Study terminated due to low accrual
Arm/Group | Treatment
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Change in Reduction of Disseminated Tumor Cells (DTC)/Mililitre (ml)
Description: Reduction of disseminated tumor cells (DTC)/ mililitre (ml) from >10DTC/ml to ≤ 10DTC/ml. DTC measured by IE/FC in patients with early stage
Time Frame: Up to 12 months
Population: Low accrual resulted in insufficient data to power statistical analyses for this outcome
Arm/Group | Treatment
Number analyzed (Participants) | 0

2. Primary Outcome: Disseminated Tumor Cell Counts
Description: Changes from baseline in disseminated tumor cell counts
Time Frame: Up to 12 months
Population: Low accrual resulted in insufficient data to power statistical analyses for this outcome
Arm/Group | Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Correlation of Local Recurrence With DTC
Description: Correlate breast cancer recurrence risk with individual values for DTC at each time point
Time Frame: Up to 12 months
Population: Low accrual resulted in insufficient data to power statistical analyses for this outcome
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=4)
cellulitis (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=4)
anxiety (Psychiatric disorders) | 1
arthralgia (Musculoskeletal and connective tissue disorders) | 1
back pain (Musculoskeletal and connective tissue disorders) | 1
breast pain (Reproductive system and breast disorders) | 1
bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
cellulitis (Skin and subcutaneous tissue disorders) | 1
elevated LFTs (Investigations) | 1
fatigue (General disorders) | 1
hypertriglyceridemia (Metabolism and nutrition disorders) | 1
lymphedema (Vascular disorders) | 1
neuroma of breast (Reproductive system and breast disorders) | 1
osteopenia (Musculoskeletal and connective tissue disorders) | 1
pain in extremity (Musculoskeletal and connective tissue disorders) | 1
syncopy episode (Nervous system disorders) | 1
vaginal discharge (Reproductive system and breast disorders) | 1
weight gain (Investigations) | 1

LIMITATIONS AND CAVEATS:
Study terminated early due to low accrual

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes